CLINICAL TRIAL: NCT01310296
Title: A Single-Center, Open-Label, Two-Period, Two-Treatment, Randomized Sequence Study to Determine the Mass Balance and Absolute Bioavailability of a Single Oral Dose of 14C-Labeled Lofexidine Compared to a Single Intravenous Dose of Lofexidine
Brief Title: Lofexidine ADME & Mass Balance in Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: USWM, LLC (dba US WorldMeds) (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: USWM-LX1-1003/ 02749MZ
Record Dates: First submitted 2011-03-04; First posted 2011-03-08 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Normal Healthy Volunteers Will be Treated With Lofexidine to Understand the Absolute Bioavailability and Mass Balance Recovery of the Product
Keywords: Phase 1; Normal Healthy Volunteers; Mass Balance; ADME; Absolute Bioavailability
MeSH Terms: interventions — lofexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiolabeled Lofexidine Oral Solution (Other): Participants will receive a radiolabeled lofexidine oral solution followed by safety evaluations, and plasma, urine and fecal sampling for up to 216 hours post dose.
  Interventions: Drug: Lofexidine hydrochloride
- Lofexidine Intravenous Solution (Experimental): Participants will receive 200 mcg of lofexidine in an intravenous solution infusion over 200 minutes followed by 72 hours of safety evaluation and plasma sampling.
  Interventions: Drug: Lofexidine hydrochloride

INTERVENTIONS:
Drug: Lofexidine hydrochloride — Single Dose = Solution containing 400 μg lofexidine HCl and a tracer amount of 14C lofexidine
  Arms: Radiolabeled Lofexidine Oral Solution
Drug: Lofexidine hydrochloride — Single Dose = 200 μg lofexidine in phosphate-buffered saline administered intravenously via infusion pump at a rate of 1 μg/min for 200 min
  Arms: Lofexidine Intravenous Solution

SUMMARY:
The purpose of this study is to determine the mass balance and absolute bioavailability of a single oral dose of 14C-labeled lofexidine compared to a single intravenous dose of lofexidine.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be a male or non-pregnant, non-breastfeeding female.
* Subject must be between 18 and 50 years of age (inclusive).
* Subject's Body Mass Index (BMI) must be between 18 and 30 kg/m2 (inclusive), and subject must weigh a minimum of 50 kg (110 lbs).
* Female subjects must agree to use one of the following forms of birth control from screening until 14 days after completion of the study:
* Vasectomized partner (at least 6 months prior to dosing)
* Post-menopausal (at least 2 years prior to dosing)
* Surgically sterile (bilateral tubal ligation, hysterectomy, bilateral oophorectomy) at least 6 months prior to dosing
* Double barrier (diaphragm with spermicide; condoms with spermicide)
* IUD (intra-uterine device)
* Abstinence (must agree to use a double barrier method if they become sexually active during the study)
* Implanted or intrauterine hormonal contraceptives in use for at least 6 consecutive months prior to study dosing and throughout the study duration
* Oral, patch, and injected contraceptives or vaginal hormonal device (i.e. NuvaRing®) in use for at least 3 consecutive months prior to study dosing and throughout the study duration.
* Subject must voluntarily consent to participate in this study and provide their written informed consent prior to start of any study- specific procedures.
* Subject is willing and able to remain in the study unit for the entire duration of each confinement period.
* Subject's vital signs must be within the following ranges to be included: Vital signs measured sitting after 3 minutes rest; heart rate: 50-90 bpm; systolic BP: 100-140 mmHg; diastolic BP: 50-90 mmHg, and oral temperature within the normal range of 35.6-37.7° C. Out-of-range vital signs may be repeated once. Predose vital signs will be assessed by the Principal Investigator or designee (e.g., a medically qualified sub-investigator) prior to study drug administration. The Principal Investigator or designee will verify the eligibility of each subject with out-of-range vital signs and document approval prior to dosing.
* For the study period in which the subject is assigned to receive Treatment A (lofexidine oral solution containing 14C-lofexidine), subject must be:
* Willing to eat entire meals and snacks provided during confinement at the research facility; and understand that the diet will include foods with high fiber content and possibly prune juice.
* Willing to remain in the clinical research center for a minimum of 7 consecutive days during pre-dose, dose, and post-dose evaluation periods. Subjects must be willing to stay for an additional 24 to 48 hours if necessary.
* Willing to collect all urine and fecal samples for the duration of the study period as required.

Exclusion Criteria:

* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.
* Has a clinically significant abnormal finding on the physical exam, medical history, ECG, or clinical laboratory results at screening.
* History of any syncopal episode or seizures.
* Presence of acute disease state (eg, nausea, vomiting, fever, diarrhea) within 7 days prior to scheduled dose administration.
* History or presence of allergic or adverse response to lofexidine or related drugs.
* Has been on a significantly abnormal diet during the 4 weeks preceding the first dose of study medication.
* Has donated blood or plasma within 30 days prior to the first dose of study medication.
* Has participated in a radiolabeled clinical trial within the last 12 months prior to the first dose of study medication.
* Has participated in another clinical trial (randomized subjects only) within 30 days prior to the first dose of study medication.
* Has used any over-the-counter (OTC) medication, including nutritional supplements, within 7 days prior to the first dose of study medication.
* Has used any prescription medication, except hormonal contraceptive or hormonal replacement therapy, within 14 days prior to the first dose of study medication.
* Subjects that have discontinued the use of implanted, intrauterine, or injected hormonal contraceptives must not have used any for 6 months prior to study start.
* Subjects that have discontinued the use of oral, patch, or vaginal hormonal contraceptives must not have used any for 1 month prior to study start.
* Has been treated with any known drugs that are moderate or strong inhibitors/inducers of CYP enzymes such as barbiturates, phenothiazines, cimetidine, carbamazepine, etc., within 30 days prior to the first dose of study medication and that in the Investigator's judgment may impact subject safety or the validity of the study results.
* Has smoked or used tobacco products within 60 days prior to the first dose of study medication.
* Has any prior history of substance abuse or treatment (including alcohol) within the past 2 years.
* Is a female with a positive pregnancy test result.
* Has a positive urine screen for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, cannabinoids, opiates).
* Has had a positive test for, or has been treated for hepatitis B, hepatitis C, or Human Immunodeficiency Virus (HIV).
* Has orthostatic hypotension at screening defined as a drop in systolic blood pressure ≥ 20 mmHg or a fall in diastolic blood pressure ≥ 10 mmHg following a 2 minute stand. Out-of-range vital signs may be repeated once. Predose vital signs will be assessed by the Principal Investigator or designee (e.g., a medically qualified sub-investigator) prior to study drug administration. The Principal Investigator or designee will verify the eligibility of each subject with out-of-range vital signs and document approval prior to dosing.
* Subjects with a QTcB greater than 450 msec (males) or greater than 470 msec (females), at screening obtained after 5 minutes rest in a supine position using the ECG machine algorithm.
* Has irregular bowel habits. ("Irregular" being defined for the purpose of this study as NOT having a bowel movement at least every 2 days.)
* Has been exposed to radiation, including dental or medical imaging such as x ray or tomography, in the 6 months prior to dose administration.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Mass Balance | plasma, urine, and fecal samples up to 216 hours post dose
  To determine the mass balance recovery of orally administered lofexidine hydrochloride

SECONDARY OUTCOMES:
Absolute Bioavailability & Tolerability | plasma samples over 72 and 144 hrs post-dose for IV and oral doses, respectively
  * To determine the absolute bioavailability of a single oral dose of lofexidine compared to a single intravenous dose of lofexidine
  * To determine the tolerability of lofexidine oral solution and intravenous lofexidine

CONTACTS AND LOCATIONS:
Overall Officials: James A Longstreth, PhD, Principal Investigator — US WorldMeds; Charles W Gorodetzky, MD, PhD, Principal Investigator — US WorldMeds; Mark Leibowitz, MD, Principal Investigator — Worldwide Clinical Trials
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States